CLINICAL TRIAL: NCT05516160
Title: Perceptually Calibrated Scale of Optical Aberrations, Generated by Multifocal Corrective Lenses
Brief Title: Perceptually Calibrated Scale of Optical Aberrations
Acronym: SOOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Collaborators: Warsaw University of Technology (Other)
Responsible Party: Principal Investigator, Karolina Krix-jachym, Principal Investigator, Military Institute od Medicine National Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 555
Record Dates: First submitted 2022-01-13; First posted 2022-08-25 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Dysphotopsia
Keywords: halo; glare; optical aberrations; multifocal lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multifocal lens (Experimental): examination of dysphotopsia
  Interventions: Diagnostic Test: diagnostic of optical aberrations
- control group (Active Comparator): examination of dysphotopsia
  Interventions: Diagnostic Test: diagnostic of optical aberrations

INTERVENTIONS:
Diagnostic Test: diagnostic of optical aberrations — diagnostic of optical aberrations with new device

SUMMARY:
The main objective of the project is to develop a new, more reliable method of modeling and parametrization of the halo and glare phenomena based on the subjective perception of these visual disturbances. The project will consist of three parts. The first will include the psychophysical measurement of glare and halo phenomena perceived by people with multifocal corrective lenses compared to the reference group. The second part will focus on the development of an algorithm for the generation of optical elements (masks) inducing standard halo and glow effects of a given size and intensity. The third phase of the project will concern the calibration of the developed algorithm. For this purpose, the halo and glare will be induced by the developed masks in the healthy eye, so as to match them with the vision disorders measured in the first part of the project in people using multifocal vision correction methods. As a result of this research, a scale for precise measurement of subjective halo and glare phenomena in the field of view will be created, independently covering their intensity and size, and in the future allowing for optical (and not graphic simulation as in commercially available simulators) simulation of scenes seen by patients.

DETAILED DESCRIPTION:
CONTENT DESCRIPTION OF THE PROJECT Perceptually calibrated scale of optical aberrations, generated by multifocal corrective lenses Scientific background:As a result of the progressive aging of the population, especially in developed countries, more and more economically active people function after cataract surgery. In Poland, approximately 250,000 patients are eligible for such a procedure annually. During it, the natural lens of the eye with a significantly limited transparency is replaced with an artificial implant, which causes the loss of eye accommodation. In order to ensure full functional vision (near, indirect and far vision), the most commonly used are implants in the form of multifocal lenses, which have become the subject of intensive research in visual optics and optometry in recent years . The search for optimal solutions to compensate for the lack of accommodation is a kind of compromise between the depth of field of view and its resolution and contrast. Often, a side effect of increasing the range of viewing distances turns out to be various types of aberrations causing distortions of the seen scenes in the form of glare and halo The glare and halo phenomena are a natural consequence of the optical properties of multifocal lenses, i.e. lenses that create two or more foci of light focus along the optical axis. Such lenses allow for sharp imaging on the screen of the retina of the eye at the same time of objects from several distances. A focused image of a point object (strictly of small angular size) placed at one of the design distances is blurred in the other. An intense bright spot (glow) appears in the center surrounded by rings of light (halo). In daytime vision, the visual centers in the human brain are shown to be good at suppressing the perception of these disturbances. The problem appears in night vision, however, when the scenes consist of light sources (lanterns, car lights, reflections) with high contrast to the background. Visible glare and halo phenomena significantly increase the threshold brightness of noticeable objects in the immediate vicinity of bright points of the field of view. Therefore, they seriously limit the safety of participation in road traffic and the comfort of vision after dark.

There are many works devoted to the problem of measuring and parametrization of the halo and glow phenomena. The first approach is based on the optical parameterization of the impulse response (PSF) and modulating transport function (MTF) of the lenses and, on their basis, the visualization of undesirable aberrations. This approach requires the use of the eye model, which is always the result of some simplifications and idealizations. It also does not take into account the physiological processes related to the vision process. Nevertheless, it allows to objectively predict the occurrence of glare and halo phenomena and associate them with a specific design of a corrective lens. It also allows to measure the size and intensity of these effects using variously defined metrics.

The second approach is to try to measure the subjective perception of halo and glow phenomena among patients with implanted or inserted multifocal lenses (Halo & Glare Simulator; Eyeland-Design Network GmbH, Vreden, Germany). Such analyzes are most often based on the method of questionnaires in which the respondents themselves determine the type of visual disturbance (from a closed graphic list) and its degree (on a quantitative scale). The task of assessing visual sensations on an interval scale is a difficult and imprecise task. Therefore, it is undoubtedly necessary to develop a more reliable, based on psychophysical methodology, quantification of the size and intensity of undesirable phenomena in the field of view.

One of the methods combining the objectivity of the study with the subjectivity of phenomena available only to the examined person is the commercially available C-quant device by Oculus (Oculus Optikgeräte, GmbH, Wetzlar, Germany), used for the diagnostic measurement of distractions in night vision. The compensatory comparison method implemented in the device consists in finding such the intensity of the flickering area located in the center of the field of view to compensate for the glow caused by the bright ring flickering in the counter-phase. With appropriately selected light intensities in the center of the field of view, the glow from the ring is visible for half a period, and a target of the same brightness for the second half of the period, so the flickering disappears. The disadvantage of this method is the result in the form of a single parameter by means of which it is impossible to precisely and independently parametrize the halo and glow phenomena.

Another method, used in the Vision Monitor device (MonCv3; Metrovision, Pérenchies, France), is a study in which the patient reads optotypes with a specific contrast placed at an increasing distance from a point light source [6]. Since the light source creates a glow and a halo in the field of view of the examined person, the minimum brightness of the identifiable individual optotypes differs depending on the distance from it. Measurement of this brightness allows to parameterize - in the analyzed device with relatively low resolution - the glow and halo phenomena in the form of their profile and intensity depending on the distance from the light source. A similar methodology will be used in the project requested for funding.

Project objectives: The main objective of the project is to develop a new, more reliable method of modeling and parametrization of the halo and glow phenomena based on the subjective perception of these visual disturbances. The project will consist of three parts. The first part will include the psychophysical measurement of glare and halo phenomena perceived by people with multifocal corrective lenses compared to the reference group. The second part will focus on the development of an algorithm for the generation of optical elements (masks) inducing standard halo and glow effects of a given size and intensity. The third phase of the project will concern the calibration of the developed algorithm. For this purpose, the halo and glare will be induced by the developed masks in the healthy eye, so as to match them with the vision disorders measured in the first part of the project in people using multifocal vision correction methods. As a result of this research, a scale for precise measurement of subjective halo and glare phenomena in the field of view will be created, independently covering their intensity and size, and in the future allowing for optical (and not graphic simulation as in commercially available simulators) simulation of scenes seen by patients.

The primary research objective of the project concerns a new method of measuring the subjective intensity and size of the halo and glow effects, as well as the construction of simple optical elements that simulate these undesirable optical phenomena in a controlled manner.

The application goal of the project is to develop a scale of optical glare and halo phenomena for use in ophthalmic diagnostics. The possibility of generating an image with the effects of glow and halo introduced in a controlled, optical way will allow in the future to design and implement devices simulating the vision of a patient using modern lenses, correcting eyesight. This will facilitate communication between the ophthalmologist and the patient both before and after cataract surgery. A continuation of this research involving a greater number of patients implanted with different multifocal lenses would probably allow linking the flare and halo effects to specific types of implants (planned public or commercialization research project). This, in turn, would enable the optimization of research into new methods of vision correction. It follows from the above that the application target has implementation potential, responding to the identified need of the medical market in the field of diagnostics of problems related to multifocal implants.

The objectives and scientific methods of the project are primarily in the areas of optical metrology and image processing included in the research plans of the Priority Research Area "Photonic Technologies". However, the project is of an interdisciplinary nature, and its potential areas of application relate to diagnostic technologies included in the research plans of POB "Biotechnoogy and Biomedical Engineering" and monitoring of the health and safety of older people included in the research plans of POB "Artificial Intelligence and Robotics".

Research methodology and plan: The research will be carried out within 24 months at the Perceptual Research Laboratory in cooperation with the Faculty of Physics and the Research and Analysis Department of the Innovation and Technology Transfer Management Center. Three research tasks and one management task will be carried out by the project manager and a team of four associates, including an ophthalmologist.

Task 1 Measurement of the field of view (4-9 month of the project) As part of the task, the recruitment of research participants will be prepared and carried out. It is planned to recruit 10 people experiencing undesirable halo and glare phenomena in the visual field as a result of using multifocal vision correction methods, and the same number of healthy people as a control group. The relatively small number of participants with implanted multifocal implants results from the fact that, unlike in the richer countries of Western Europe, cataract surgery with multifocal lenses is not so common in Poland, due to the lack of reimbursement from the National Health Fund. Nevertheless, the current project should be treated as a pilot project in order to apply for funds for extensive clinical trials on the developed solutions. The basic test will be the measurement of the field of view (perimetry) in simulated night conditions in the presence of a strong, point light source in the central field. The visibility of additional weak point light sources, appropriately distributed in the field of view, should be significantly disturbed by the effects of flash and halo. Researchers expect that a detailed analysis of the field of view in such conditions will allow us to determine the spatial perceptual characteristics of the field of view in the form of a map of the threshold light intensity detected by the examined person at particular points of the field of view. In turn, on the basis of such a map, it wille be possible to determine the angular dimensions and intensity distribution, corresponding to the perceived effects of glow and halo. Examination of the field of view of participants from the control group will be used to reliably verify whether the results obtained in the case of people after cataract surgery are clearly related to the implantation of multifocal implants.

Task 2. Construction of an algorithm for the generation of optical elements and simulation of their operation (10-15 month of the project) The main goal of the task will be to develop an algorithm that generates model halo and glow phenomena. The task will involve preparing optical elements (masks) generating images of points in the form of a spot simulating the glow effect and a concentric ring around this spot simulating the halo effect. The developed algorithm will be based on the generation of Bessel and Gauss beams and the controlled shaping of the light beam. The parameters of the elements will be calibrated using psychophysical methodology in such a way that the induced phenomena correspond to the disturbances experienced by patients. Patients will independently define the size, relative intensity of the spot and the ring, and will become a quantitative measure of the corresponding halo and glare effects in subjective vision.

Task 3. Perceptual calibration of the developed scale. (16-21 month of the project) The primary goal of the task will be perceptual calibration of the created pattern optical effects. For this purpose, it will be verified whether the flash phenomena and halos perceived as a result of using multifocal lenses can be reliably reproduced (with the same parameters) in people from the control group. The research will be carried out in a vision simulator, constructed as part of the independently implemented project "VIDO - improving vision with the help of dynamic optics" (LIDER / 15/0061 / L-9/17 / NCBR / 2018, implementation period 2019-2021). The vision simulator enables the study of visual perception after correction of the optical system of the eye with any computer-generated optical elements and placed virtually in the entrance pupil of the eye. The parameters of the disturbance-generating elements will be adjusted to those perceived by people with multifocal lenses. A quantitative measure of perceived halo and glow phenomena will be possible.

Task 4. Project management (1-24 month of the project) Project management will be based on elements of the PRINCE2 methodology. The task consists of three steps. In the first (1-3 month) project initiation will be carried out, consisting in submitting an application to the bioethics committee, establishing a strategy for delegating tasks, the flow of their documentation, quality control and progress in their implementation, as well as a strategy for controlling and reporting risks related to the project implementation. Purchases of the necessary materials and equipment will also be commissioned, as well as prepared contracts with project contractors. The second stage of the task (4-21 months) will be the ongoing coordination and control of the performance of tasks in accordance with the principles and criteria set out in the adopted strategies. The final stage will be project closure (month 22-24). As part of this phase of the task implementation, the assumptions adopted in the project plan will be compared with the results achieved, reports on the project implementation will be prepared, and publications on the project results will be prepared and submitted.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females, of any race
* one or both eyes with implanted intraocular monofocal lens (10 eyes) and multifocal lens (10 eyes)
* informed consent to participate in the study
* presence at scheduled follow-up visits after the procedure for a period of 24 months.

Exclusion Criteria:

* in the eye qualified for the test:

  * cataract
  * Fuchs dystrophy and other corneal diseases
  * evidence of serious eye disease
  * ophthalmic surgeries other than cataract surgery
  * clinically active or past uveitis
  * intraocular pressure (IOP) >21 mmHg
  * glaucoma
  * retinal detachment or its suspicion in ultrasound examination of the eyeball
  * systemic diseases with ocular symptoms, including diseases that may affect the function of corneal endothelial cells
* intolerance of the examination in the slit lamp or other procedures planned in the examination
* pregnancy
* mental disorders or emotional instability to an extent that does not allow the subject's informed consent in the study and presence at scheduled follow-up visits
* documented sensitivity to pharmacological agents used in the study, i.e. topical anesthetics, fluorescein, other related to the ophthalmological examination serious fatal illnesses or a patient's medical condition preventing the study from continuing for a period of 6 months
* current participation in other research programs
* therapy with oral anticoagulants

the participant may withdraw from the study at any time and for any reason without consequences and without prohibiting participation in other research projects. A participant may not return to the current study again if he or she has previously withdrawn.

Termination of participation in the study may take place in the case of:

1. decrease in visual acuity >3 Snellen lines from baseline (> 15 letters ETDRS, >0.3 logMAR) in one of the eyes
2. the presence of adverse symptoms or complications associated or not with the examination, which affect the ability to see or the functioning of the body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-09 (Estimated); Primary Completion 2022-12-29 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
presence of optical aberrations in analyzed eyes | up to 3 months
  halo and glare presence in analyzed eyes

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Krix-Jachym, MD PhD, Principal Investigator — Military Institute of Warsaw, Poland

REFERENCES:
- [Background] Song X, Liu X, Wang W, Zhu Y, Qin Z, Lyu D, Shentu X, Xv W, Chen P, Ke Y. Visual outcome and optical quality after implantation of zonal refractive multifocal and extended-range-of-vision IOLs: a prospective comparison. J Cataract Refract Surg. 2020 Apr;46(4):540-548. doi: 10.1097/j.jcrs.0000000000000088. PMID 32213781
- [Background] Carson D, Lee S, Alexander E, Wei X, Lee S. Comparison of two laboratory-based systems for evaluation of halos in intraocular lenses. Clin Ophthalmol. 2018 Feb 21;12:385-393. doi: 10.2147/OPTH.S152201. eCollection 2018. PMID 29503526
- [Background] Savini G, Schiano-Lomoriello D, Balducci N, Barboni P. Visual Performance of a New Extended Depth-of-Focus Intraocular Lens Compared to a Distance-Dominant Diffractive Multifocal Intraocular Lens. J Refract Surg. 2018 Apr 1;34(4):228-235. doi: 10.3928/1081597X-20180125-01. PMID 29634837